CLINICAL TRIAL: NCT04293354
Title: Analgesic Efficacy of Serratus Anterior Plane Block in The Rib Fractures Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Gözen Öksüz, associate professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/11-18
Record Dates: First submitted 2020-02-29; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Serratus Plane Block

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus Plane Block (Active Comparator): The Serratus plane block was performed, tramadol was administered with patient-controlled analgesia (PCA) and all patients were followed in the ward.
  Interventions: Procedure: Serratus Plane Block
- Control (Sham Comparator): No block was performed, tramadol was administered with patient-controlled analgesia (PCA) and all patients were followed in the ward.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Serratus Plane Block — Serratus Plane Block was performed
  Arms: Serratus Plane Block
Procedure: Control — No block was performed
  Arms: Control

SUMMARY:
Serratus Anterior Plane Block (SAPB) is a facial plane block that was first described by Blanco in 2013 and that blocks the lateral cutaneous branches of the T2-T9 intercostal nerves, the intercostobrachial nerve, n. thoracic longus, n. thoracodorsalis nerves. Case and case series have been reported in the literature on the use of SAPB in rib fractures, and it has been reported as an effective analgesia method. We apply SAPB to patients with rib fractures with pain in our clinic.

Our aim is to evaluate SAPB for patients with rib fractures pain and to compare them with the control group in terms of total analgesic consumption and pain scores.

DETAILED DESCRIPTION:
After Ethics Committee approval patients with rib fracture pain and have a Numerical Rating Scale (NRS) score of ≥ 4, included the study. The patients were randomized by the closed envelope method. The patients were divided into two groups as the SAPB-performed group (Group S) and the Control group (Group K). Intravenous patient-controlled analgesia (PCA) device prepared with tramadol was applied to all patients.

ELIGIBILITY:
Inclusion Criteria:

Rib fracture pain and had a Numerical Rating Scale (NRS) score of ≥ 4 ASA I-II-III

Exclusion Criteria:

Patients with infection at the injection site Coagulopathy Allergy to amide-type local anesthetics History of peripheral neuropathy Hepatic and/or renal failure Refusing the procedure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Analgesic consumption | up to 24 hour
  Tramadol

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) | at 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 12 hours, 24 hours
  pain scores

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras Sutcu Imam University Hospital, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Okmen K, Okmen BM. The efficacy of serratus anterior plane block in analgesia for thoracotomy: a retrospective study. J Anesth. 2017 Aug;31(4):579-585. doi: 10.1007/s00540-017-2364-9. Epub 2017 Apr 26. PMID 28447227
- [Derived] Teksen S, Oksuz G, Oksuz H, Sayan M, Arslan M, Urfalioglu A, Gisi G, Bilal B. Analgesic efficacy of the serratus anterior plane block in rib fractures pain: A randomized controlled trial. Am J Emerg Med. 2021 Mar;41:16-20. doi: 10.1016/j.ajem.2020.12.041. Epub 2020 Dec 23. PMID 33383266